CLINICAL TRIAL: NCT00886288
Title: A Comparison of Telmisartan Effectiveness in Hypertensive Patients With and Without Albuminuria.
Brief Title: TELMA - Observational Study in Daily Medical Practice of the Effectiveness of Telmisartan for Treatment of Hypertension in Patients With and Without Confirmed Albuminuria in Belgium
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.521
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2009-11-18 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Telmisartan
- Telmisartan + hydrochlorothiazide

SUMMARY:
This study was carried out in the context of daily medical practice to compare the effectiveness of telmisartan in the treatment of hypertension complicated or not with the presence of protein in the urine, which is called albuminuria. Hypertension is a chronic, treatable but not curable disease and is defined as a combination of a systolic blood pressure of 140 mmHg or more and a diastolic pressure of 90 mmHg or more. The kidneys are often the first organs damaged by hypertension; renal damage could easily be diagnosed using a urine dipstick and should be part of a routine examination in hypertensive patient. The aim of the study is to see if the decrease of blood pressure (both systolic and diastolic) after approximately 12 weeks of treatment with telmisartan in patients with albuminuria is the same or different to that in patients without albuminuria. Every patient participating should have two visits, approximately 12 weeks apart where his/her blood pressure was checked and a few questions about is concomitant disease and drugs were asked.

ELIGIBILITY:
Inclusion criteria:

Age above or equal to 18, no upper limit Patient has been treated and followed up for more than 6 months by the same general practitioner (GP) Hypertension treated for at least 3 months and not under control at the time of inclusion in the study [systolic blood pressure (SBP) above or equal to 140 mmHg and diastolic blood pressure (DBP) above or equal to 90 mmHg, or SBP above or equal to 130 mmHg and DBP above or equal to 80 mmHg if patient has chronic renal insufficiency or diabetes] Results available from at least two tests of albuminuria Antihypertensive treatment remained unchanged during the month prior data collection Decision by the GP to introduce telmisartan (either in combination with hydrochlorthiazide [HCTZ] or not) in the antihypertensive treatment (normal prescription) Written informed consent of the patient to collect his/her data

Exclusion criteria:

Blood pressure under control [SBP below 140 mmHg and DBP below 90 mmHg or SBP below 130 mmHg and DBP below 80 mmHg if patient has chronic renal insufficiency or diabetes] The patient refuse to allow his/her data to be collected Women of childbearing potential not using an effective contraception method, as well as women who are breastfeeding Patients with proteinuria above or equal to 1g/l or with glomerular filtration rate (GFR) below 15 ml/min/1.73 m² Current or prior use of telmisartan within the last 12 months Change in the antihypertensive treatment during the month prior to collection of the data

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients
Sampling Method: Probability Sample
Enrollment: 2874 (Actual)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (936):
- Belgium (936):
  - Boehringer Ingelheim Investigational Site 1, Aalst
  - Boehringer Ingelheim Investigational Site 2, Aalst
  - Boehringer Ingelheim Investigational Site 3, Aalst
  - Boehringer Ingelheim Investigational Site 4, Aalst
  - Boehringer Ingelheim Investigational Site 5, Aalter
  - Boehringer Ingelheim Investigational Site 6, Aalter
  - Boehringer Ingelheim Investigational Site 10, Aarschot
  - Boehringer Ingelheim Investigational Site 11, Aarschot
  - Boehringer Ingelheim Investigational Site 7, Aarschot
  - Boehringer Ingelheim Investigational Site 8, Aarschot
  - Boehringer Ingelheim Investigational Site 9, Aarschot
  - Boehringer Ingelheim Investigational Site 12, Adinkerke
  - Boehringer Ingelheim Investigational Site 13, Affligem
  - Boehringer Ingelheim Investigational Site 14, Affligem-Hekeigem
  - Boehringer Ingelheim Investigational Site 15, Alleur
  - Boehringer Ingelheim Investigational Site 16, Alleur
  - Boehringer Ingelheim Investigational Site 17, Alleur
  - Boehringer Ingelheim Investigational Site 18, Alleur
  - Boehringer Ingelheim Investigational Site 19, Alveringem
  - Boehringer Ingelheim Investigational Site 20, Amay
  - Boehringer Ingelheim Investigational Site 21, Amay
  - Boehringer Ingelheim Investigational Site 22, Amougies
  - Boehringer Ingelheim Investigational Site 23, Anderlues
  - Boehringer Ingelheim Investigational Site 24, Anderlues
  - Boehringer Ingelheim Investigational Site 25, Angleur
  - Boehringer Ingelheim Investigational Site 26, Ans
  - Boehringer Ingelheim Investigational Site 27, Ans
  - Boehringer Ingelheim Investigational Site 28, Ans
  - Boehringer Ingelheim Investigational Site 29, Ans
  - Boehringer Ingelheim Investigational Site 30, Ans
  - Boehringer Ingelheim Investigational Site 31, Anthisnes
  - Boehringer Ingelheim Investigational Site 32, Antoing
  - Boehringer Ingelheim Investigational Site 33, Antwerp
  - Boehringer Ingelheim Investigational Site 34, Antwerp
  - Boehringer Ingelheim Investigational Site 35, Antwerp
  - Boehringer Ingelheim Investigational Site 36, Anzegem
  - Boehringer Ingelheim Investigational Site 37, Anzegem
  - Boehringer Ingelheim Investigational Site 38, Arquennes
  - Boehringer Ingelheim Investigational Site 39, Asquillies
  - Boehringer Ingelheim Investigational Site 40, Asse
  - Boehringer Ingelheim Investigational Site 41, Asse
  - Boehringer Ingelheim Investigational Site 42, Ath
  - Boehringer Ingelheim Investigational Site 43, Auvelais
  - Boehringer Ingelheim Investigational Site 44, Awans
  - Boehringer Ingelheim Investigational Site 45, Awans
  - Boehringer Ingelheim Investigational Site 46, Ayeneux
  - Boehringer Ingelheim Investigational Site 47, Baardegem
  - Boehringer Ingelheim Investigational Site 48, Baasrode
  - Boehringer Ingelheim Investigational Site 49, Basècles
  - Boehringer Ingelheim Investigational Site 50, Bassilly
  - Boehringer Ingelheim Investigational Site 51, Battice
  - Boehringer Ingelheim Investigational Site 52, Bazel
  - Boehringer Ingelheim Investigational Site 53, Beaufays
  - Boehringer Ingelheim Investigational Site 54, Beaufays-Chaudfontaine
  - Boehringer Ingelheim Investigational Site 55, Beauraing
  - Boehringer Ingelheim Investigational Site 56, Beauraing
  - Boehringer Ingelheim Investigational Site 57, Beernem
  - Boehringer Ingelheim Investigational Site 58, Beerzel
  - Boehringer Ingelheim Investigational Site 59, Begijnendijk
  - Boehringer Ingelheim Investigational Site 60, Belgrade
  - Boehringer Ingelheim Investigational Site 61, Belgrade
  - Boehringer Ingelheim Investigational Site 62, Belgrade
  - Boehringer Ingelheim Investigational Site 63, Bellaire
  - Boehringer Ingelheim Investigational Site 64, Belsele
  - Boehringer Ingelheim Investigational Site 65, Belzele
  - Boehringer Ingelheim Investigational Site 66, Ben-Ahin
  - Boehringer Ingelheim Investigational Site 67, Beringen
  - Boehringer Ingelheim Investigational Site 68, Beringen
  - Boehringer Ingelheim Investigational Site 69, Berlaar
  - Boehringer Ingelheim Investigational Site 70, Bertrix
  - Boehringer Ingelheim Investigational Site 71, Betekom
  - Boehringer Ingelheim Investigational Site 72, Betekom
  - Boehringer Ingelheim Investigational Site 73, Beveren
  - Boehringer Ingelheim Investigational Site 74, Beverlo
  - Boehringer Ingelheim Investigational Site 75, Beverlo
  - Boehringer Ingelheim Investigational Site 76, Beverlo
  - Boehringer Ingelheim Investigational Site 77, Beverlo
  - Boehringer Ingelheim Investigational Site 78, Beyne-Heusay
  - Boehringer Ingelheim Investigational Site 79, Beyne-Heusay
  - Boehringer Ingelheim Investigational Site 80, Beyne-Heusay
  - Boehringer Ingelheim Investigational Site 81, Beyne-Heusay
  - Boehringer Ingelheim Investigational Site 82, Bierghes-Rebecq
  - Boehringer Ingelheim Investigational Site 83, Bilstain
  - Boehringer Ingelheim Investigational Site 84, Bilzen
  - Boehringer Ingelheim Investigational Site 85, Bilzen
  - Boehringer Ingelheim Investigational Site 86, Bilzen
  - Boehringer Ingelheim Investigational Site 87, Bilzen
  - Boehringer Ingelheim Investigational Site 88, Bilzen
  - Boehringer Ingelheim Investigational Site 89, Binche
  - Boehringer Ingelheim Investigational Site 90, Binche
  - Boehringer Ingelheim Investigational Site 91, Binche
  - Boehringer Ingelheim Investigational Site 92, Binche
  - Boehringer Ingelheim Investigational Site 93, Blaregnies
  - Boehringer Ingelheim Investigational Site 94, Blaton
  - Boehringer Ingelheim Investigational Site 95, Blégny
  - Boehringer Ingelheim Investigational Site 96, Boezinge
  - Boehringer Ingelheim Investigational Site 97, Bois de Villiers
  - Boehringer Ingelheim Investigational Site 100, Bois-d'Haine
  - Boehringer Ingelheim Investigational Site 99, Bois-d'Haine
  - Boehringer Ingelheim Investigational Site 98, Bois-de-Villers
  - Boehringer Ingelheim Investigational Site 101, Boncelles
  - Boehringer Ingelheim Investigational Site 102, Boncelles
  - Boehringer Ingelheim Investigational Site 103, Boolschot
  - Boehringer Ingelheim Investigational Site 104, Boolschot
  - Boehringer Ingelheim Investigational Site 105, Borgerhout
  - Boehringer Ingelheim Investigational Site 106, Bornem
  - Boehringer Ingelheim Investigational Site 107, Bornem
  - Boehringer Ingelheim Investigational Site 108, Bornem
  - Boehringer Ingelheim Investigational Site 109, Bornem
  - Boehringer Ingelheim Investigational Site 110, Bouffioulx
  - Boehringer Ingelheim Investigational Site 111, Bouillon
  - Boehringer Ingelheim Investigational Site 112, Bouillon
  - Boehringer Ingelheim Investigational Site 113, Boussu
  - Boehringer Ingelheim Investigational Site 114, Boussu
  - Boehringer Ingelheim Investigational Site 115, Braine-l'Alleud
  - Boehringer Ingelheim Investigational Site 116, Braine-l'Alleud
  - Boehringer Ingelheim Investigational Site 117, Braine-l'Alleud
  - Boehringer Ingelheim Investigational Site 118, Braine-l'Alleud
  - Boehringer Ingelheim Investigational Site 119, Braine-l'Alleud
  - Boehringer Ingelheim Investigational Site 120, Braine-l'Alleud
  - Boehringer Ingelheim Investigational Site 121, Braine-le-Château
  - Boehringer Ingelheim Investigational Site 122, Braine-le-Château
  - Boehringer Ingelheim Investigational Site 123, Braine-le-Comte
  - Boehringer Ingelheim Investigational Site 124, Brakel
  - Boehringer Ingelheim Investigational Site 125, Brakel
  - Boehringer Ingelheim Investigational Site 126, Brakel
  - Boehringer Ingelheim Investigational Site 127, Brasschaat
  - Boehringer Ingelheim Investigational Site 128, Brasschaat
  - Boehringer Ingelheim Investigational Site 129, Brasschaat
  - Boehringer Ingelheim Investigational Site 130, Brasschaat
  - Boehringer Ingelheim Investigational Site 131, Brasschaat
  - Boehringer Ingelheim Investigational Site 132, Brasschaat
  - Boehringer Ingelheim Investigational Site 133, Brasschaat
  - Boehringer Ingelheim Investigational Site 134, Bray
  - Boehringer Ingelheim Investigational Site 135, Brecht
  - Boehringer Ingelheim Investigational Site 136, Brecht
  - Boehringer Ingelheim Investigational Site 137, Brecht
  - Boehringer Ingelheim Investigational Site 138, Brecht
  - Boehringer Ingelheim Investigational Site 139, Bredene
  - Boehringer Ingelheim Investigational Site 140, Bree
  - Boehringer Ingelheim Investigational Site 141, Bree
  - Boehringer Ingelheim Investigational Site 142, Bruges
  - Boehringer Ingelheim Investigational Site 143, Bruges
  - Boehringer Ingelheim Investigational Site 144, Bruges
  - Boehringer Ingelheim Investigational Site 145, Bruges
  - Boehringer Ingelheim Investigational Site 146, Bruges
  - Boehringer Ingelheim Investigational Site 147, Bruges
  - Boehringer Ingelheim Investigational Site 148, Bruges
  - Boehringer Ingelheim Investigational Site 149, Bruges
  - Boehringer Ingelheim Investigational Site 150, Brussels
  - Boehringer Ingelheim Investigational Site 151, Brussels
  - Boehringer Ingelheim Investigational Site 152, Brussels
  - Boehringer Ingelheim Investigational Site 153, Brussels
  - Boehringer Ingelheim Investigational Site 154, Brussels
  - Boehringer Ingelheim Investigational Site 155, Brussels
  - Boehringer Ingelheim Investigational Site 156, Brussels
  - Boehringer Ingelheim Investigational Site 157, Brussels
  - Boehringer Ingelheim Investigational Site 158, Brussels
  - Boehringer Ingelheim Investigational Site 159, Brussels
  - Boehringer Ingelheim Investigational Site 160, Brussels
  - Boehringer Ingelheim Investigational Site 161, Brussels
  - Boehringer Ingelheim Investigational Site 162, Brussels
  - Boehringer Ingelheim Investigational Site 163, Brussels
  - Boehringer Ingelheim Investigational Site 164, Brussels
  - Boehringer Ingelheim Investigational Site 165, Brussels
  - Boehringer Ingelheim Investigational Site 166, Brussels
  - Boehringer Ingelheim Investigational Site 167, Brussels
  - Boehringer Ingelheim Investigational Site 168, Brussels
  - Boehringer Ingelheim Investigational Site 169, Brussels
  - Boehringer Ingelheim Investigational Site 170, Brussels
  - Boehringer Ingelheim Investigational Site 171, Brussels
  - Boehringer Ingelheim Investigational Site 172, Brussels
  - Boehringer Ingelheim Investigational Site 173, Brussels
  - Boehringer Ingelheim Investigational Site 174, Brussels
  - Boehringer Ingelheim Investigational Site 175, Brussels
  - Boehringer Ingelheim Investigational Site 176, Brussels
  - Boehringer Ingelheim Investigational Site 177, Brussels
  - Boehringer Ingelheim Investigational Site 178, Brussels
  - Boehringer Ingelheim Investigational Site 179, Brussels
  - Boehringer Ingelheim Investigational Site 180, Brussels
  - Boehringer Ingelheim Investigational Site 181, Brussels
  - Boehringer Ingelheim Investigational Site 182, Brussels
  - Boehringer Ingelheim Investigational Site 183, Brussels
  - Boehringer Ingelheim Investigational Site 184, Brussels
  - Boehringer Ingelheim Investigational Site 185, Brussels
  - Boehringer Ingelheim Investigational Site 186, Brussels
  - Boehringer Ingelheim Investigational Site 187, Brussels
  - Boehringer Ingelheim Investigational Site 188, Brussels
  - Boehringer Ingelheim Investigational Site 189, Brussels
  - Boehringer Ingelheim Investigational Site 190, Brussels
  - Boehringer Ingelheim Investigational Site 191, Brussels
  - Boehringer Ingelheim Investigational Site 192, Brussels
  - Boehringer Ingelheim Investigational Site 193, Brussels
  - Boehringer Ingelheim Investigational Site 194, Brussels
  - Boehringer Ingelheim Investigational Site 195, Brussels
  - Boehringer Ingelheim Investigational Site 196, Brussels
  - Boehringer Ingelheim Investigational Site 197, Brussels
  - Boehringer Ingelheim Investigational Site 198, Brussels
  - Boehringer Ingelheim Investigational Site 199, Brussels
  - Boehringer Ingelheim Investigational Site 200, Brussels
  - Boehringer Ingelheim Investigational Site 201, Brussels
  - Boehringer Ingelheim Investigational Site 202, Brussels
  - Boehringer Ingelheim Investigational Site 203, Brussels
  - Boehringer Ingelheim Investigational Site 204, Brussels
  - Boehringer Ingelheim Investigational Site 205, Brussels
  - Boehringer Ingelheim Investigational Site 206, Brussels
  - Boehringer Ingelheim Investigational Site 207, Brussels
  - Boehringer Ingelheim Investigational Site 208, Brussels
  - Boehringer Ingelheim Investigational Site 209, Brussels
  - Boehringer Ingelheim Investigational Site 210, Brussels
  - Boehringer Ingelheim Investigational Site 211, Brussels
  - Boehringer Ingelheim Investigational Site 212, Brussels
  - Boehringer Ingelheim Investigational Site 213, Buizingen
  - Boehringer Ingelheim Investigational Site 214, Burcht
  - Boehringer Ingelheim Investigational Site 215, Burdinne
  - Boehringer Ingelheim Investigational Site 216, Burst
  - Boehringer Ingelheim Investigational Site 217, Buvrinnes
  - Boehringer Ingelheim Investigational Site 218, Carnières
  - Boehringer Ingelheim Investigational Site 219, Carnières
  - Boehringer Ingelheim Investigational Site 220, Charleroi
  - Boehringer Ingelheim Investigational Site 221, Châtelineau
  - Boehringer Ingelheim Investigational Site 222, Chênée
  - Boehringer Ingelheim Investigational Site 223, Chièvres
  - Boehringer Ingelheim Investigational Site 224, Ciney
  - Boehringer Ingelheim Investigational Site 225, Ciney
  - Boehringer Ingelheim Investigational Site 226, Clavier
  - Boehringer Ingelheim Investigational Site 227, Colfontaine
  - Boehringer Ingelheim Investigational Site 228, Court-St-Etienne
  - Boehringer Ingelheim Investigational Site 229, Dalhem
  - Boehringer Ingelheim Investigational Site 230, De Haan
  - Boehringer Ingelheim Investigational Site 231, De Pinte
  - Boehringer Ingelheim Investigational Site 232, De Pinte
  - Boehringer Ingelheim Investigational Site 233, De Pinte
  - Boehringer Ingelheim Investigational Site 234, Deinze
  - Boehringer Ingelheim Investigational Site 235, Deinze
  - Boehringer Ingelheim Investigational Site 236, Deinze
  - Boehringer Ingelheim Investigational Site 237, Den Haan Aan Zee
  - Boehringer Ingelheim Investigational Site 238, Denderhoutem
  - Boehringer Ingelheim Investigational Site 239, Denderhoutem
  - Boehringer Ingelheim Investigational Site 240, Denderhoutem
  - Boehringer Ingelheim Investigational Site 241, Denderleeuw
  - Boehringer Ingelheim Investigational Site 242, Dessel
  - Boehringer Ingelheim Investigational Site 243, Deurne
  - Boehringer Ingelheim Investigational Site 244, Deurne
  - Boehringer Ingelheim Investigational Site 245, Deurne
  - Boehringer Ingelheim Investigational Site 246, Deurne
  - Boehringer Ingelheim Investigational Site 247, Deurne
  - Boehringer Ingelheim Investigational Site 248, Deux-Acrem-Lessines
  - Boehringer Ingelheim Investigational Site 249, Diepenbeek
  - Boehringer Ingelheim Investigational Site 250, Diepenbeek
  - Boehringer Ingelheim Investigational Site 251, Diest
  - Boehringer Ingelheim Investigational Site 252, Diest
  - Boehringer Ingelheim Investigational Site 253, Dikkebus
  - Boehringer Ingelheim Investigational Site 254, Diksmuide
  - Boehringer Ingelheim Investigational Site 255, Dilbeek
  - Boehringer Ingelheim Investigational Site 256, Dilbeek
  - Boehringer Ingelheim Investigational Site 257, Dion-Valmont
  - Boehringer Ingelheim Investigational Site 258, Doische
  - Boehringer Ingelheim Investigational Site 259, Dottignies
  - Boehringer Ingelheim Investigational Site 260, Dour
  - Boehringer Ingelheim Investigational Site 261, Drogenbos
  - Boehringer Ingelheim Investigational Site 262, Drongen
  - Boehringer Ingelheim Investigational Site 263, Duffel
  - Boehringer Ingelheim Investigational Site 264, Duffel
  - Boehringer Ingelheim Investigational Site 265, Dworp
  - Boehringer Ingelheim Investigational Site 266, Ecaussines
  - Boehringer Ingelheim Investigational Site 267, Ecaussines
  - Boehringer Ingelheim Investigational Site 268, Ecaussines
  - Boehringer Ingelheim Investigational Site 269, Edegem
  - Boehringer Ingelheim Investigational Site 270, Edegem
  - Boehringer Ingelheim Investigational Site 271, Edegem
  - Boehringer Ingelheim Investigational Site 272, Eeklo
  - Boehringer Ingelheim Investigational Site 273, Eeklo
  - Boehringer Ingelheim Investigational Site 274, Eernegem
  - Boehringer Ingelheim Investigational Site 275, Ekeren
  - Boehringer Ingelheim Investigational Site 276, Enghien
  - Boehringer Ingelheim Investigational Site 277, Engis
  - Boehringer Ingelheim Investigational Site 278, Ensival
  - Boehringer Ingelheim Investigational Site 279, Erembodegem
  - Boehringer Ingelheim Investigational Site 280, Eremnodegem
  - Boehringer Ingelheim Investigational Site 281, Erpe
  - Boehringer Ingelheim Investigational Site 282, Erpe
  - Boehringer Ingelheim Investigational Site 283, Erpe-Mere
  - Boehringer Ingelheim Investigational Site 284, Erpe-Mere
  - Boehringer Ingelheim Investigational Site 285, Erpe-Mere
  - Boehringer Ingelheim Investigational Site 286, Erpe-Mere
  - Boehringer Ingelheim Investigational Site 287, Erpent
  - Boehringer Ingelheim Investigational Site 288, Escanaffles
  - Boehringer Ingelheim Investigational Site 289, Essen
  - Boehringer Ingelheim Investigational Site 290, Essen
  - Boehringer Ingelheim Investigational Site 291, Eupen
  - Boehringer Ingelheim Investigational Site 292, Eupen
  - Boehringer Ingelheim Investigational Site 293, Eupen
  - Boehringer Ingelheim Investigational Site 294, Evegnée
  - Boehringer Ingelheim Investigational Site 295, Fairon
  - Boehringer Ingelheim Investigational Site 296, Feluy
  - Boehringer Ingelheim Investigational Site 297, Flawinne
  - Boehringer Ingelheim Investigational Site 298, Flawinne
  - Boehringer Ingelheim Investigational Site 304, Fleurus
  - Boehringer Ingelheim Investigational Site 305, Fleurus
  - Boehringer Ingelheim Investigational Site 299, Flémalle
  - Boehringer Ingelheim Investigational Site 300, Flémalle
  - Boehringer Ingelheim Investigational Site 301, Flémalle
  - Boehringer Ingelheim Investigational Site 302, Flémalle
  - Boehringer Ingelheim Investigational Site 303, Flémalle
  - Boehringer Ingelheim Investigational Site 306, Florenville
  - Boehringer Ingelheim Investigational Site 307, Fosses-la-Ville
  - Boehringer Ingelheim Investigational Site 308, Frameries
  - Boehringer Ingelheim Investigational Site 309, Francorchamps
  - Boehringer Ingelheim Investigational Site 310, Frasnes
  - Boehringer Ingelheim Investigational Site 311, Frasnes
  - Boehringer Ingelheim Investigational Site 312, Galmaarden
  - Boehringer Ingelheim Investigational Site 313, Geel
  - Boehringer Ingelheim Investigational Site 314, Geel
  - Boehringer Ingelheim Investigational Site 315, Geel
  - Boehringer Ingelheim Investigational Site 316, Geel
  - Boehringer Ingelheim Investigational Site 317, Gembloux
  - Boehringer Ingelheim Investigational Site 318, Gembloux
  - Boehringer Ingelheim Investigational Site 319, Genk
  - Boehringer Ingelheim Investigational Site 320, Genk
  - Boehringer Ingelheim Investigational Site 321, Genk
  - Boehringer Ingelheim Investigational Site 322, Genk
  - Boehringer Ingelheim Investigational Site 323, Genk
  - Boehringer Ingelheim Investigational Site 324, Genk
  - Boehringer Ingelheim Investigational Site 325, Genk
  - Boehringer Ingelheim Investigational Site 326, Genk
  - Boehringer Ingelheim Investigational Site 327, Genk
  - Boehringer Ingelheim Investigational Site 332, Gentbrugge
  - Boehringer Ingelheim Investigational Site 333, Genval
  - Boehringer Ingelheim Investigational Site 334, Geraardsbergen
  - Boehringer Ingelheim Investigational Site 335, Gerpinnes
  - Boehringer Ingelheim Investigational Site 328, Ghent
  - Boehringer Ingelheim Investigational Site 329, Ghent
  - Boehringer Ingelheim Investigational Site 330, Ghent
  - Boehringer Ingelheim Investigational Site 331, Ghent
  - Boehringer Ingelheim Investigational Site 336, Ghlin
  - Boehringer Ingelheim Investigational Site 337, Gijzegem
  - Boehringer Ingelheim Investigational Site 338, Gingelom
  - Boehringer Ingelheim Investigational Site 339, Gingelon
  - Boehringer Ingelheim Investigational Site 340, Gits
  - Boehringer Ingelheim Investigational Site 341, Givry
  - Boehringer Ingelheim Investigational Site 532, Glain
  - Boehringer Ingelheim Investigational Site 342, Gooik
  - Boehringer Ingelheim Investigational Site 343, Gooreind-Wuustwezel
  - Boehringer Ingelheim Investigational Site 344, Gozée
  - Boehringer Ingelheim Investigational Site 345, Gozée
  - Boehringer Ingelheim Investigational Site 346, Grâce-Hollogne
  - Boehringer Ingelheim Investigational Site 347, Grâce-Hollogne
  - Boehringer Ingelheim Investigational Site 348, Grez-Doiceau
  - Boehringer Ingelheim Investigational Site 349, Grimbergen
  - Boehringer Ingelheim Investigational Site 350, Grimbergen
  - Boehringer Ingelheim Investigational Site 351, Grimbergen
  - Boehringer Ingelheim Investigational Site 352, Grimminge
  - Boehringer Ingelheim Investigational Site 353, Grivegnée
  - Boehringer Ingelheim Investigational Site 354, Grivegnée
  - Boehringer Ingelheim Investigational Site 355, Grobbendonk
  - Boehringer Ingelheim Investigational Site 356, Grobbendonk
  - Boehringer Ingelheim Investigational Site 357, Groot Bijgarden
  - Boehringer Ingelheim Investigational Site 358, Gruitrode
  - Boehringer Ingelheim Investigational Site 359, Gullegem
  - Boehringer Ingelheim Investigational Site 360, Haaltert
  - Boehringer Ingelheim Investigational Site 361, Haaltert
  - Boehringer Ingelheim Investigational Site 362, Halen
  - Boehringer Ingelheim Investigational Site 363, Halen
  - Boehringer Ingelheim Investigational Site 364, Halle
  - Boehringer Ingelheim Investigational Site 365, Halle
  - Boehringer Ingelheim Investigational Site 366, Halle
  - Boehringer Ingelheim Investigational Site 367, Halle
  - Boehringer Ingelheim Investigational Site 368, Halle
  - Boehringer Ingelheim Investigational Site 369, Ham
  - Boehringer Ingelheim Investigational Site 370, Hamme
  - Boehringer Ingelheim Investigational Site 371, Hamme
  - Boehringer Ingelheim Investigational Site 372, Hamme
  - Boehringer Ingelheim Investigational Site 373, Hamoir
  - Boehringer Ingelheim Investigational Site 374, Hamoir
  - Boehringer Ingelheim Investigational Site 375, Harelbeke
  - Boehringer Ingelheim Investigational Site 376, Hasselt
  - Boehringer Ingelheim Investigational Site 377, Hasselt
  - Boehringer Ingelheim Investigational Site 378, Havay
  - Boehringer Ingelheim Investigational Site 379, Heist-op-den-Berg
  - Boehringer Ingelheim Investigational Site 380, Heist-op-den-Berg
  - Boehringer Ingelheim Investigational Site 381, Hellebecq
  - Boehringer Ingelheim Investigational Site 383, Hemiksem
  - Boehringer Ingelheim Investigational Site 382, Hemikse
  - Boehringer Ingelheim Investigational Site 384, Heppen-Leopoldsburg
  - Boehringer Ingelheim Investigational Site 385, Herseaux
  - Boehringer Ingelheim Investigational Site 386, Herselt
  - Boehringer Ingelheim Investigational Site 387, Herselt
  - Boehringer Ingelheim Investigational Site 388, Herselt
  - Boehringer Ingelheim Investigational Site 389, Herstal
  - Boehringer Ingelheim Investigational Site 390, Herstal
  - Boehringer Ingelheim Investigational Site 391, Herzele
  - Boehringer Ingelheim Investigational Site 392, Herzele
  - Boehringer Ingelheim Investigational Site 393, Herzele
  - Boehringer Ingelheim Investigational Site 394, Herzele
  - Boehringer Ingelheim Investigational Site 395, Herzele
  - Boehringer Ingelheim Investigational Site 396, Heusden-Zolder
  - Boehringer Ingelheim Investigational Site 397, Heusy
  - Boehringer Ingelheim Investigational Site 398, Hever
  - Boehringer Ingelheim Investigational Site 399, Heverlee
  - Boehringer Ingelheim Investigational Site 400, Heverlee
  - Boehringer Ingelheim Investigational Site 401, Hoboken
  - Boehringer Ingelheim Investigational Site 402, Hoboken
  - Boehringer Ingelheim Investigational Site 403, Hoeilaart
  - Boehringer Ingelheim Investigational Site 404, Hoeilaart
  - Boehringer Ingelheim Investigational Site 405, Hoeselt
  - Boehringer Ingelheim Investigational Site 406, Hoeselt
  - Boehringer Ingelheim Investigational Site 407, Hofstade-Aalst
  - Boehringer Ingelheim Investigational Site 408, Hognoul
  - Boehringer Ingelheim Investigational Site 409, Hollogne-sur-Geer
  - Boehringer Ingelheim Investigational Site 410, Hombeek
  - Boehringer Ingelheim Investigational Site 411, Hooglede
  - Boehringer Ingelheim Investigational Site 412, Hooglede
  - Boehringer Ingelheim Investigational Site 413, Hornu
  - Boehringer Ingelheim Investigational Site 414, Hornu
  - Boehringer Ingelheim Investigational Site 415, Hotton
  - Boehringer Ingelheim Investigational Site 416, Houdeng-Aimeries
  - Boehringer Ingelheim Investigational Site 417, Houdeng-Aimeries
  - Boehringer Ingelheim Investigational Site 418, Houdeng-Aimeries
  - Boehringer Ingelheim Investigational Site 419, Houdeng-Goegnies
  - Boehringer Ingelheim Investigational Site 420, Houthalen
  - Boehringer Ingelheim Investigational Site 421, Houthalen
  - Boehringer Ingelheim Investigational Site 422, Houthalen
  - Boehringer Ingelheim Investigational Site 423, Houthulst-Klerken
  - Boehringer Ingelheim Investigational Site 424, Houtvenne
  - Boehringer Ingelheim Investigational Site 425, Houyet
  - Boehringer Ingelheim Investigational Site 426, Hove
  - Boehringer Ingelheim Investigational Site 427, Hove
  - Boehringer Ingelheim Investigational Site 428, Huy
  - Boehringer Ingelheim Investigational Site 429, Huy
  - Boehringer Ingelheim Investigational Site 430, Ichtegem
  - Boehringer Ingelheim Investigational Site 431, Ieper
  - Boehringer Ingelheim Investigational Site 432, Ieper
  - Boehringer Ingelheim Investigational Site 433, Ingelmunster
  - Boehringer Ingelheim Investigational Site 434, Ingelmunster
  - Boehringer Ingelheim Investigational Site 435, Ingelmunster
  - Boehringer Ingelheim Investigational Site 436, Ingelmunster
  - Boehringer Ingelheim Investigational Site 437, Itegem
  - Boehringer Ingelheim Investigational Site 438, Itegem
  - Boehringer Ingelheim Investigational Site 439, Itterbeek
  - Boehringer Ingelheim Investigational Site 440, Izegem
  - Boehringer Ingelheim Investigational Site 441, Izegem
  - Boehringer Ingelheim Investigational Site 442, Izegem
  - Boehringer Ingelheim Investigational Site 443, Izegem
  - Boehringer Ingelheim Investigational Site 444, Izegem
  - Boehringer Ingelheim Investigational Site 445, Jabbeke
  - Boehringer Ingelheim Investigational Site 446, Jalhay
  - Boehringer Ingelheim Investigational Site 447, Jambes
  - Boehringer Ingelheim Investigational Site 448, Jambes
  - Boehringer Ingelheim Investigational Site 449, Jemappes
  - Boehringer Ingelheim Investigational Site 451, Jemeppe-Seraing
  - Boehringer Ingelheim Investigational Site 450, Jemeppe-sur-Sambre
  - Boehringer Ingelheim Investigational Site 452, Jollain
  - Boehringer Ingelheim Investigational Site 453, Jumet
  - Boehringer Ingelheim Investigational Site 454, Jumet
  - Boehringer Ingelheim Investigational Site 455, Jumet
  - Boehringer Ingelheim Investigational Site 456, Jupille Liège
  - Boehringer Ingelheim Investigational Site 457, Juprelle
  - Boehringer Ingelheim Investigational Site 458, Kachten-Izegem
  - Boehringer Ingelheim Investigational Site 459, Kain
  - Boehringer Ingelheim Investigational Site 460, Kalken
  - Boehringer Ingelheim Investigational Site 461, Kapelle O/d Bos
  - Boehringer Ingelheim Investigational Site 462, Kapellen
  - Boehringer Ingelheim Investigational Site 463, Kaprijke
  - Boehringer Ingelheim Investigational Site 464, Kasterbee
  - Boehringer Ingelheim Investigational Site 465, Kessel-Lo
  - Boehringer Ingelheim Investigational Site 466, Kessel-Lo
  - Boehringer Ingelheim Investigational Site 467, Kettenis
  - Boehringer Ingelheim Investigational Site 468, Kieldrecht
  - Boehringer Ingelheim Investigational Site 469, Knesselare
  - Boehringer Ingelheim Investigational Site 470, Knokke
  - Boehringer Ingelheim Investigational Site 471, Knokke-Heist
  - Boehringer Ingelheim Investigational Site 472, Knokke-Heist
  - Boehringer Ingelheim Investigational Site 473, Koekelare
  - Boehringer Ingelheim Investigational Site 474, Koekelare
  - Boehringer Ingelheim Investigational Site 475, Koningshooikt
  - Boehringer Ingelheim Investigational Site 476, Kontich
  - Boehringer Ingelheim Investigational Site 477, Kontich
  - Boehringer Ingelheim Investigational Site 478, Kortemark
  - Boehringer Ingelheim Investigational Site 479, Kortemark
  - Boehringer Ingelheim Investigational Site 481, Kortijk-Dutsel
  - Boehringer Ingelheim Investigational Site 480, Kortijk
  - Boehringer Ingelheim Investigational Site 482, Kortrijk
  - Boehringer Ingelheim Investigational Site 483, Kortrijk
  - Boehringer Ingelheim Investigational Site 484, Kortrijk
  - Boehringer Ingelheim Investigational Site 485, Kortrijk - Aalbeke
  - Boehringer Ingelheim Investigational Site 486, Kortrijk-Dutsel
  - Boehringer Ingelheim Investigational Site 487, Kraainem
  - Boehringer Ingelheim Investigational Site 488, Kraainem
  - Boehringer Ingelheim Investigational Site 489, Kruishoutem
  - Boehringer Ingelheim Investigational Site 490, Kuringen
  - Boehringer Ingelheim Investigational Site 491, Kuurne
  - Boehringer Ingelheim Investigational Site 492, La Boulerie
  - Boehringer Ingelheim Investigational Site 493, La Bouverie
  - Boehringer Ingelheim Investigational Site 494, La Hestre
  - Boehringer Ingelheim Investigational Site 495, La Louvière
  - Boehringer Ingelheim Investigational Site 496, La Reid
  - Boehringer Ingelheim Investigational Site 497, Laakdal
  - Boehringer Ingelheim Investigational Site 498, Laarne
  - Boehringer Ingelheim Investigational Site 499, Langeark
  - Boehringer Ingelheim Investigational Site 500, Lauwe
  - Boehringer Ingelheim Investigational Site 501, Lavacherie
  - Boehringer Ingelheim Investigational Site 502, Lede
  - Boehringer Ingelheim Investigational Site 503, Ledegem
  - Boehringer Ingelheim Investigational Site 504, Ledegem
  - Boehringer Ingelheim Investigational Site 505, Ledegem
  - Boehringer Ingelheim Investigational Site 506, Ledegem
  - Boehringer Ingelheim Investigational Site 507, Leefdaal
  - Boehringer Ingelheim Investigational Site 508, Leers-et-Fosteau
  - Boehringer Ingelheim Investigational Site 509, Lembeek
  - Boehringer Ingelheim Investigational Site 510, Lens
  - Boehringer Ingelheim Investigational Site 511, Leopoldsburg
  - Boehringer Ingelheim Investigational Site 512, Leopoldsburg
  - Boehringer Ingelheim Investigational Site 513, Lessines
  - Boehringer Ingelheim Investigational Site 514, Lessines
  - Boehringer Ingelheim Investigational Site 515, Lessines
  - Boehringer Ingelheim Investigational Site 516, Leut-Maasmechelen
  - Boehringer Ingelheim Investigational Site 517, Leuven
  - Boehringer Ingelheim Investigational Site 518, Leuven
  - Boehringer Ingelheim Investigational Site 519, Leuven
  - Boehringer Ingelheim Investigational Site 520, Leuven
  - Boehringer Ingelheim Investigational Site 521, Leuven
  - Boehringer Ingelheim Investigational Site 522, Leuze En Hainaut
  - Boehringer Ingelheim Investigational Site 523, Libin
  - Boehringer Ingelheim Investigational Site 524, Libramont
  - Boehringer Ingelheim Investigational Site 525, Lichtervelde
  - Boehringer Ingelheim Investigational Site 533, Lier
  - Boehringer Ingelheim Investigational Site 534, Lier
  - Boehringer Ingelheim Investigational Site 526, Liège
  - Boehringer Ingelheim Investigational Site 527, Liège
  - Boehringer Ingelheim Investigational Site 528, Liège
  - Boehringer Ingelheim Investigational Site 529, Liège
  - Boehringer Ingelheim Investigational Site 530, Liège
  - Boehringer Ingelheim Investigational Site 531, Liège
  - Boehringer Ingelheim Investigational Site 535, Lint
  - Boehringer Ingelheim Investigational Site 536, Linter
  - Boehringer Ingelheim Investigational Site 545, Lo-Reninge
  - Boehringer Ingelheim Investigational Site 546, Lo-Reninge
  - Boehringer Ingelheim Investigational Site 537, Lobbes
  - Boehringer Ingelheim Investigational Site 538, Lochristi
  - Boehringer Ingelheim Investigational Site 539, Lochristi
  - Boehringer Ingelheim Investigational Site 540, Lokeren
  - Boehringer Ingelheim Investigational Site 541, Lokeren
  - Boehringer Ingelheim Investigational Site 542, Lokeren
  - Boehringer Ingelheim Investigational Site 543, Lokeren
  - Boehringer Ingelheim Investigational Site 544, Lokeren
  - Boehringer Ingelheim Investigational Site 547, Loupoigne
  - Boehringer Ingelheim Investigational Site 548, Louveigné
  - Boehringer Ingelheim Investigational Site 549, Lovendegem
  - Boehringer Ingelheim Investigational Site 550, Luingne
  - Boehringer Ingelheim Investigational Site 551, Luttre
  - Boehringer Ingelheim Investigational Site 552, Maasmechelen
  - Boehringer Ingelheim Investigational Site 553, Manhay
  - Boehringer Ingelheim Investigational Site 554, Marche
  - Boehringer Ingelheim Investigational Site 555, Marche-en-Famenne
  - Boehringer Ingelheim Investigational Site 556, Marche-en-Famenne
  - Boehringer Ingelheim Investigational Site 557, Marloie
  - Boehringer Ingelheim Investigational Site 558, Marloie
  - Boehringer Ingelheim Investigational Site 559, Massenhoven
  - Boehringer Ingelheim Investigational Site 560, Massenhoven
  - Boehringer Ingelheim Investigational Site 561, Mechelen
  - Boehringer Ingelheim Investigational Site 562, Mechelen
  - Boehringer Ingelheim Investigational Site 563, Mechelen
  - Boehringer Ingelheim Investigational Site 564, Mechelen
  - Boehringer Ingelheim Investigational Site 565, Mechelen
  - Boehringer Ingelheim Investigational Site 566, Meerhout
  - Boehringer Ingelheim Investigational Site 567, Meerhout
  - Boehringer Ingelheim Investigational Site 568, Meerhout
  - Boehringer Ingelheim Investigational Site 569, Meerhout
  - Boehringer Ingelheim Investigational Site 571, Menen
  - Boehringer Ingelheim Investigational Site 572, Menen
  - Boehringer Ingelheim Investigational Site 573, Mere
  - Boehringer Ingelheim Investigational Site 574, Merkem
  - Boehringer Ingelheim Investigational Site 575, Merksem
  - Boehringer Ingelheim Investigational Site 576, Merksem
  - Boehringer Ingelheim Investigational Site 577, Merlebeke
  - Boehringer Ingelheim Investigational Site 578, Meslin L'evèque
  - Boehringer Ingelheim Investigational Site 579, Messelbroek
  - Boehringer Ingelheim Investigational Site 580, Mettet
  - Boehringer Ingelheim Investigational Site 581, Mettet
  - Boehringer Ingelheim Investigational Site 582, Mettet
  - Boehringer Ingelheim Investigational Site 583, Meux
  - Boehringer Ingelheim Investigational Site 570, Mélin
  - Boehringer Ingelheim Investigational Site 584, Middekerke
  - Boehringer Ingelheim Investigational Site 585, Middelkerke
  - Boehringer Ingelheim Investigational Site 586, Mignault
  - Boehringer Ingelheim Investigational Site 587, Modauf
  - Boehringer Ingelheim Investigational Site 588, Moerbeke-Waas
  - Boehringer Ingelheim Investigational Site 589, Moerzeke
  - Boehringer Ingelheim Investigational Site 590, Moha (Wanze)
  - Boehringer Ingelheim Investigational Site 591, Mol
  - Boehringer Ingelheim Investigational Site 592, Mol
  - Boehringer Ingelheim Investigational Site 593, Mol
  - Boehringer Ingelheim Investigational Site 594, Mol
  - Boehringer Ingelheim Investigational Site 595, Mons
  - Boehringer Ingelheim Investigational Site 600, Mont-St-Aubert
  - Boehringer Ingelheim Investigational Site 601, Mont-St-Aubert
  - Boehringer Ingelheim Investigational Site 596, Montenaken
  - Boehringer Ingelheim Investigational Site 597, Montignies-sur-Sambre
  - Boehringer Ingelheim Investigational Site 598, Montignies-sur-Sambre
  - Boehringer Ingelheim Investigational Site 599, Montigny-Tilleul
  - Boehringer Ingelheim Investigational Site 602, Montzen
  - Boehringer Ingelheim Investigational Site 603, Moorsel
  - Boehringer Ingelheim Investigational Site 604, Moorsel
  - Boehringer Ingelheim Investigational Site 609, Morlanwelz-Carnières
  - Boehringer Ingelheim Investigational Site 605, Morlanwelz-Mariemont
  - Boehringer Ingelheim Investigational Site 606, Morlanwelz-Mariemont
  - Boehringer Ingelheim Investigational Site 607, Morlanwelz-Mariemont
  - Boehringer Ingelheim Investigational Site 608, Morlanwelz-Mariemont
  - Boehringer Ingelheim Investigational Site 610, Mortsel
  - Boehringer Ingelheim Investigational Site 611, Mouscron
  - Boehringer Ingelheim Investigational Site 612, Mouscron
  - Boehringer Ingelheim Investigational Site 613, Mouscron
  - Boehringer Ingelheim Investigational Site 614, Mouscron
  - Boehringer Ingelheim Investigational Site 615, Mouscron
  - Boehringer Ingelheim Investigational Site 616, Mouscron
  - Boehringer Ingelheim Investigational Site 617, Mouscron
  - Boehringer Ingelheim Investigational Site 618, Muizen
  - Boehringer Ingelheim Investigational Site 619, Namur
  - Boehringer Ingelheim Investigational Site 620, Namur
  - Boehringer Ingelheim Investigational Site 621, Namur
  - Boehringer Ingelheim Investigational Site 622, Namur
  - Boehringer Ingelheim Investigational Site 623, Naninne
  - Boehringer Ingelheim Investigational Site 624, Natoye
  - Boehringer Ingelheim Investigational Site 625, Neerlinder
  - Boehringer Ingelheim Investigational Site 626, Neerpelt
  - Boehringer Ingelheim Investigational Site 627, Neufvilles
  - Boehringer Ingelheim Investigational Site 628, Nieuwkerke
  - Boehringer Ingelheim Investigational Site 629, Ninove
  - Boehringer Ingelheim Investigational Site 630, Ninove
  - Boehringer Ingelheim Investigational Site 631, Ninove
  - Boehringer Ingelheim Investigational Site 632, Nismes
  - Boehringer Ingelheim Investigational Site 633, Nivelles
  - Boehringer Ingelheim Investigational Site 634, Nivelles
  - Boehringer Ingelheim Investigational Site 635, Nivelles
  - Boehringer Ingelheim Investigational Site 636, Nivelles
  - Boehringer Ingelheim Investigational Site 637, Noorderwijk
  - Boehringer Ingelheim Investigational Site 638, Olen
  - Boehringer Ingelheim Investigational Site 639, Olen
  - Boehringer Ingelheim Investigational Site 640, Olen
  - Boehringer Ingelheim Investigational Site 641, Olmen-Balen
  - Boehringer Ingelheim Investigational Site 642, Olmen-Balen
  - Boehringer Ingelheim Investigational Site 649, Oostham-Ham
  - Boehringer Ingelheim Investigational Site 650, Oostkamp
  - Boehringer Ingelheim Investigational Site 651, Oostnieuwkerke
  - Boehringer Ingelheim Investigational Site 652, Oostrozebeke
  - Boehringer Ingelheim Investigational Site 802, Oplinter
  - Boehringer Ingelheim Investigational Site 653, Oreye
  - Boehringer Ingelheim Investigational Site 643, Ostend
  - Boehringer Ingelheim Investigational Site 644, Ostend
  - Boehringer Ingelheim Investigational Site 645, Ostend
  - Boehringer Ingelheim Investigational Site 646, Ostend
  - Boehringer Ingelheim Investigational Site 647, Ostend
  - Boehringer Ingelheim Investigational Site 648, Ostend
  - Boehringer Ingelheim Investigational Site 654, Otegem
  - Boehringer Ingelheim Investigational Site 655, Othée
  - Boehringer Ingelheim Investigational Site 656, Ottignies
  - Boehringer Ingelheim Investigational Site 661, Oud-Turnhout
  - Boehringer Ingelheim Investigational Site 662, Oud-Turnhout
  - Boehringer Ingelheim Investigational Site 657, Oudegem
  - Boehringer Ingelheim Investigational Site 658, Oudenaarde
  - Boehringer Ingelheim Investigational Site 659, Oudenaarde
  - Boehringer Ingelheim Investigational Site 660, Oudenaarde
  - Boehringer Ingelheim Investigational Site 663, Ougrée
  - Boehringer Ingelheim Investigational Site 664, Outer
  - Boehringer Ingelheim Investigational Site 665, Overijse
  - Boehringer Ingelheim Investigational Site 666, Overpelt
  - Boehringer Ingelheim Investigational Site 667, Passendale
  - Boehringer Ingelheim Investigational Site 668, Pepinster
  - Boehringer Ingelheim Investigational Site 669, Perllaines
  - Boehringer Ingelheim Investigational Site 671, Petit-Rechain
  - Boehringer Ingelheim Investigational Site 670, Péronnes
  - Boehringer Ingelheim Investigational Site 672, Philippeville
  - Boehringer Ingelheim Investigational Site 673, Piéton
  - Boehringer Ingelheim Investigational Site 674, Piéton
  - Boehringer Ingelheim Investigational Site 675, Pittem
  - Boehringer Ingelheim Investigational Site 676, Poederlee
  - Boehringer Ingelheim Investigational Site 677, Poederlee
  - Boehringer Ingelheim Investigational Site 678, Poelkapelle
  - Boehringer Ingelheim Investigational Site 679, Poelkappelle
  - Boehringer Ingelheim Investigational Site 680, Pondrôme
  - Boehringer Ingelheim Investigational Site 681, Poperinge
  - Boehringer Ingelheim Investigational Site 682, Posses-La-Ville
  - Boehringer Ingelheim Investigational Site 683, Pottes
  - Boehringer Ingelheim Investigational Site 684, Profondeville
  - Boehringer Ingelheim Investigational Site 685, Puurs
  - Boehringer Ingelheim Investigational Site 686, Puurs
  - Boehringer Ingelheim Investigational Site 687, Quevaucamps
  - Boehringer Ingelheim Investigational Site 688, Quevy
  - Boehringer Ingelheim Investigational Site 689, Raeren
  - Boehringer Ingelheim Investigational Site 690, Ransart
  - Boehringer Ingelheim Investigational Site 691, Ransart
  - Boehringer Ingelheim Investigational Site 692, Rendeux
  - Boehringer Ingelheim Investigational Site 693, Ressaix
  - Boehringer Ingelheim Investigational Site 694, Rijkevorsel
  - Boehringer Ingelheim Investigational Site 695, Rijkevorsel
  - Boehringer Ingelheim Investigational Site 696, Rillaar
  - Boehringer Ingelheim Investigational Site 697, Rillaar
  - Boehringer Ingelheim Investigational Site 698, Rixensart
  - Boehringer Ingelheim Investigational Site 699, Rixensart
  - Boehringer Ingelheim Investigational Site 700, Robertville
  - Boehringer Ingelheim Investigational Site 701, Rochefort
  - Boehringer Ingelheim Investigational Site 702, Roeselaar
  - Boehringer Ingelheim Investigational Site 703, Roeselaar
  - Boehringer Ingelheim Investigational Site 704, Roeselare - Oekene
  - Boehringer Ingelheim Investigational Site 705, Roeslare
  - Boehringer Ingelheim Investigational Site 706, Roeslare
  - Boehringer Ingelheim Investigational Site 707, Roeslare
  - Boehringer Ingelheim Investigational Site 708, Roloux
  - Boehringer Ingelheim Investigational Site 709, Ronquières
  - Boehringer Ingelheim Investigational Site 710, Ronse
  - Boehringer Ingelheim Investigational Site 711, Roosdaal
  - Boehringer Ingelheim Investigational Site 712, Roosdaal
  - Boehringer Ingelheim Investigational Site 713, Rotselaar
  - Boehringer Ingelheim Investigational Site 714, Rotselaar
  - Boehringer Ingelheim Investigational Site 715, Ruisbroek
  - Boehringer Ingelheim Investigational Site 716, Ruisbroek
  - Boehringer Ingelheim Investigational Site 717, Rummen
  - Boehringer Ingelheim Investigational Site 718, Rupelmonde
  - Boehringer Ingelheim Investigational Site 767, Saint Truiden
  - Boehringer Ingelheim Investigational Site 722, Saint-Denis
  - Boehringer Ingelheim Investigational Site 765, Saint-Denis
  - Boehringer Ingelheim Investigational Site 766, Saint-Denis
  - Boehringer Ingelheim Investigational Site 773, Saint-Hubert
  - Boehringer Ingelheim Investigational Site 719, Saint-Vaast
  - Boehringer Ingelheim Investigational Site 720, Saint-Vaast
  - Boehringer Ingelheim Investigational Site 721, Saint-Vaast
  - Boehringer Ingelheim Investigational Site 724, Saive
  - Boehringer Ingelheim Investigational Site 725, Sambreville
  - Boehringer Ingelheim Investigational Site 723, Sankt Vith
  - Boehringer Ingelheim Investigational Site 782, Sankt Vith
  - Boehringer Ingelheim Investigational Site 726, Sart-Bernard
  - Boehringer Ingelheim Investigational Site 727, Schendelbeke
  - Boehringer Ingelheim Investigational Site 728, Scherpenheuvel
  - Boehringer Ingelheim Investigational Site 729, Schiplaken
  - Boehringer Ingelheim Investigational Site 730, Schoten
  - Boehringer Ingelheim Investigational Site 731, Seraing
  - Boehringer Ingelheim Investigational Site 732, Seraing
  - Boehringer Ingelheim Investigational Site 733, Sinaai
  - Boehringer Ingelheim Investigational Site 734, Sint-Amands
  - Boehringer Ingelheim Investigational Site 735, Sint-Amandsberg
  - Boehringer Ingelheim Investigational Site 736, Sint-Amandsberg
  - Boehringer Ingelheim Investigational Site 737, Sint-Amandsberg
  - Boehringer Ingelheim Investigational Site 738, Sint-Denijs-Westrem
  - Boehringer Ingelheim Investigational Site 739, Sint-Genesius-Rode
  - Boehringer Ingelheim Investigational Site 740, Sint-Genesius-Rode
  - Boehringer Ingelheim Investigational Site 741, Sint-Job-In't-Goor
  - Boehringer Ingelheim Investigational Site 742, Sint-Niklaas
  - Boehringer Ingelheim Investigational Site 743, Sint-Niklaas
  - Boehringer Ingelheim Investigational Site 744, Sint-Niklaas
  - Boehringer Ingelheim Investigational Site 745, Sint-Niklaas
  - Boehringer Ingelheim Investigational Site 746, Sint-Niklaas
  - Boehringer Ingelheim Investigational Site 747, Sint-Niklaas
  - Boehringer Ingelheim Investigational Site 748, Sint-Pieters-Leeuw
  - Boehringer Ingelheim Investigational Site 749, Sint-Pieters-Leeuw
  - Boehringer Ingelheim Investigational Site 750, Sint-Truiden
  - Boehringer Ingelheim Investigational Site 751, Sivry-Rance
  - Boehringer Ingelheim Investigational Site 752, Slijpe
  - Boehringer Ingelheim Investigational Site 753, Soignies
  - Boehringer Ingelheim Investigational Site 754, Somme-Leuze
  - Boehringer Ingelheim Investigational Site 755, Soumagne
  - Boehringer Ingelheim Investigational Site 756, Sovet
  - Boehringer Ingelheim Investigational Site 757, Spa
  - Boehringer Ingelheim Investigational Site 758, Spa
  - Boehringer Ingelheim Investigational Site 759, Spa
  - Boehringer Ingelheim Investigational Site 760, Spirmont
  - Boehringer Ingelheim Investigational Site 761, Spontin
  - Boehringer Ingelheim Investigational Site 762, Sprimont
  - Boehringer Ingelheim Investigational Site 763, Spy
  - Boehringer Ingelheim Investigational Site 764, Spy
  - Boehringer Ingelheim Investigational Site 772, St-Gillis
  - Boehringer Ingelheim Investigational Site 774, St-Kat-Waver
  - Boehringer Ingelheim Investigational Site 775, St-L-Houtem
  - Boehringer Ingelheim Investigational Site 776, St-Niklaas
  - Boehringer Ingelheim Investigational Site 777, St-Niklaas
  - Boehringer Ingelheim Investigational Site 778, St-Niklaas
  - Boehringer Ingelheim Investigational Site 779, St-Pauwels
  - Boehringer Ingelheim Investigational Site 781, St-Truiden
  - Boehringer Ingelheim Investigational Site 768, Stabroek
  - Boehringer Ingelheim Investigational Site 769, Stambruges
  - Boehringer Ingelheim Investigational Site 770, Stavelot
  - Boehringer Ingelheim Investigational Site 771, Stembert
  - Boehringer Ingelheim Investigational Site 780, Strépy-Bracquegnies
  - Boehringer Ingelheim Investigational Site 783, Taintignies
  - Boehringer Ingelheim Investigational Site 784, Tamines
  - Boehringer Ingelheim Investigational Site 785, Temse
  - Boehringer Ingelheim Investigational Site 786, Terhagen
  - Boehringer Ingelheim Investigational Site 787, Ternat
  - Boehringer Ingelheim Investigational Site 788, Tessenderlo
  - Boehringer Ingelheim Investigational Site 789, Tessenderlo
  - Boehringer Ingelheim Investigational Site 790, Tessenderlo
  - Boehringer Ingelheim Investigational Site 791, Tessenderlo
  - Boehringer Ingelheim Investigational Site 792, Tessenderlo
  - Boehringer Ingelheim Investigational Site 793, Tessenderlo
  - Boehringer Ingelheim Investigational Site 794, Testelt
  - Boehringer Ingelheim Investigational Site 795, Theux
  - Boehringer Ingelheim Investigational Site 796, Theux
  - Boehringer Ingelheim Investigational Site 797, Thiméon
  - Boehringer Ingelheim Investigational Site 798, Thy-Le-Baudouin
  - Boehringer Ingelheim Investigational Site 799, Tielt
  - Boehringer Ingelheim Investigational Site 800, Tienen
  - Boehringer Ingelheim Investigational Site 801, Tienen
  - Boehringer Ingelheim Investigational Site 803, Tilleur
  - Boehringer Ingelheim Investigational Site 804, Tisselt
  - Boehringer Ingelheim Investigational Site 805, Tongeren
  - Boehringer Ingelheim Investigational Site 806, Tongeren
  - Boehringer Ingelheim Investigational Site 807, Tongeren
  - Boehringer Ingelheim Investigational Site 808, Tongeren
  - Boehringer Ingelheim Investigational Site 809, Torhout
  - Boehringer Ingelheim Investigational Site 810, Torhout
  - Boehringer Ingelheim Investigational Site 811, Tournai
  - Boehringer Ingelheim Investigational Site 812, Tournai
  - Boehringer Ingelheim Investigational Site 813, Trivières
  - Boehringer Ingelheim Investigational Site 814, Trois-Ponts
  - Boehringer Ingelheim Investigational Site 815, Trois-Ponts
  - Boehringer Ingelheim Investigational Site 816, Tubize
  - Boehringer Ingelheim Investigational Site 817, Tubize
  - Boehringer Ingelheim Investigational Site 818, Tubize
  - Boehringer Ingelheim Investigational Site 819, Tubize
  - Boehringer Ingelheim Investigational Site 820, Tubize-Oisquercq
  - Boehringer Ingelheim Investigational Site 821, Turnhout
  - Boehringer Ingelheim Investigational Site 822, Turnhout
  - Boehringer Ingelheim Investigational Site 823, Uccle
  - Boehringer Ingelheim Investigational Site 824, Uccle
  - Boehringer Ingelheim Investigational Site 825, Varsenare - Jabbeke
  - Boehringer Ingelheim Investigational Site 826, Vaux-sur-Sûre
  - Boehringer Ingelheim Investigational Site 827, Veerle
  - Boehringer Ingelheim Investigational Site 828, Velm
  - Boehringer Ingelheim Investigational Site 829, Velm
  - Boehringer Ingelheim Investigational Site 830, Verlaine
  - Boehringer Ingelheim Investigational Site 831, Verviers
  - Boehringer Ingelheim Investigational Site 832, Verviers
  - Boehringer Ingelheim Investigational Site 833, Verviers
  - Boehringer Ingelheim Investigational Site 834, Verviers
  - Boehringer Ingelheim Investigational Site 835, Verviers
  - Boehringer Ingelheim Investigational Site 836, Verviers
  - Boehringer Ingelheim Investigational Site 837, Verviers
  - Boehringer Ingelheim Investigational Site 838, Verviers
  - Boehringer Ingelheim Investigational Site 839, Verviers
  - Boehringer Ingelheim Investigational Site 840, Vezon
  - Boehringer Ingelheim Investigational Site 841, Viane
  - Boehringer Ingelheim Investigational Site 842, Vielsam
  - Boehringer Ingelheim Investigational Site 843, Villers-Poterie
  - Boehringer Ingelheim Investigational Site 844, Villiers-le-Bouillet
  - Boehringer Ingelheim Investigational Site 845, Villiers-le-Temple
  - Boehringer Ingelheim Investigational Site 846, Vinderhoute
  - Boehringer Ingelheim Investigational Site 847, Vissenaken
  - Boehringer Ingelheim Investigational Site 848, Vitrival
  - Boehringer Ingelheim Investigational Site 849, Vlezenbeek/St P.L.
  - Boehringer Ingelheim Investigational Site 850, Vlinmenen
  - Boehringer Ingelheim Investigational Site 851, Voeren-Fournon
  - Boehringer Ingelheim Investigational Site 852, Voorde
  - Boehringer Ingelheim Investigational Site 853, Vorselaar
  - Boehringer Ingelheim Investigational Site 854, Vosselaar
  - Boehringer Ingelheim Investigational Site 855, Vosselaar
  - Boehringer Ingelheim Investigational Site 856, Vrasene
  - Boehringer Ingelheim Investigational Site 857, Waarschoot
  - Boehringer Ingelheim Investigational Site 858, Waasmunter
  - Boehringer Ingelheim Investigational Site 859, Wagnelée
  - Boehringer Ingelheim Investigational Site 860, Waha
  - Boehringer Ingelheim Investigational Site 861, Waimes
  - Boehringer Ingelheim Investigational Site 862, Wambeek
  - Boehringer Ingelheim Investigational Site 863, Wanze
  - Boehringer Ingelheim Investigational Site 864, Wanze
  - Boehringer Ingelheim Investigational Site 865, Wanze
  - Boehringer Ingelheim Investigational Site 866, Waregem
  - Boehringer Ingelheim Investigational Site 867, Waregem
  - Boehringer Ingelheim Investigational Site 868, Waterloo
  - Boehringer Ingelheim Investigational Site 869, Waterloo
  - Boehringer Ingelheim Investigational Site 870, Waterloo
  - Boehringer Ingelheim Investigational Site 871, Waterloo
  - Boehringer Ingelheim Investigational Site 872, Watermael-Boitsfort
  - Boehringer Ingelheim Investigational Site 873, Watou
  - Boehringer Ingelheim Investigational Site 874, Wavre
  - Boehringer Ingelheim Investigational Site 875, Wavre
  - Boehringer Ingelheim Investigational Site 876, Wavre
  - Boehringer Ingelheim Investigational Site 877, Wavreille
  - Boehringer Ingelheim Investigational Site 878, Welkenraedt
  - Boehringer Ingelheim Investigational Site 879, Welkenraedt
  - Boehringer Ingelheim Investigational Site 880, Welle
  - Boehringer Ingelheim Investigational Site 881, Wellin
  - Boehringer Ingelheim Investigational Site 882, Wellin
  - Boehringer Ingelheim Investigational Site 883, Welvelgem
  - Boehringer Ingelheim Investigational Site 884, Werbomont
  - Boehringer Ingelheim Investigational Site 885, Wervik
  - Boehringer Ingelheim Investigational Site 886, Westende
  - Boehringer Ingelheim Investigational Site 887, Westerlo
  - Boehringer Ingelheim Investigational Site 888, Westerlo
  - Boehringer Ingelheim Investigational Site 889, Westmeerbeek
  - Boehringer Ingelheim Investigational Site 890, Westmeerbeek
  - Boehringer Ingelheim Investigational Site 891, Westrozebeke
  - Boehringer Ingelheim Investigational Site 892, Wetteren
  - Boehringer Ingelheim Investigational Site 893, Wetteren
  - Boehringer Ingelheim Investigational Site 894, Wetteren
  - Boehringer Ingelheim Investigational Site 895, Wevelgem
  - Boehringer Ingelheim Investigational Site 896, Wichelen
  - Boehringer Ingelheim Investigational Site 897, Wiekevorst
  - Boehringer Ingelheim Investigational Site 898, Wijnegem
  - Boehringer Ingelheim Investigational Site 899, Wijnegem
  - Boehringer Ingelheim Investigational Site 900, Wijnegem
  - Boehringer Ingelheim Investigational Site 901, Wijnegem
  - Boehringer Ingelheim Investigational Site 902, Wijnegem
  - Boehringer Ingelheim Investigational Site 903, Willebroek
  - Boehringer Ingelheim Investigational Site 904, Willebroek
  - Boehringer Ingelheim Investigational Site 905, Willebroek
  - Boehringer Ingelheim Investigational Site 906, Wilrijk
  - Boehringer Ingelheim Investigational Site 907, Wilryk
  - Boehringer Ingelheim Investigational Site 908, Wingene
  - Boehringer Ingelheim Investigational Site 909, Woluwé Saint-Lambert
  - Boehringer Ingelheim Investigational Site 910, Woumen
  - Boehringer Ingelheim Investigational Site 911, Woustwezel
  - Boehringer Ingelheim Investigational Site 912, Wuustwezel
  - Boehringer Ingelheim Investigational Site 913, Xhoris
  - Boehringer Ingelheim Investigational Site 914, Xhoris
  - Boehringer Ingelheim Investigational Site 915, Zarren
  - Boehringer Ingelheim Investigational Site 916, Zedelgem
  - Boehringer Ingelheim Investigational Site 917, Zeebrugge
  - Boehringer Ingelheim Investigational Site 918, Zeldegem
  - Boehringer Ingelheim Investigational Site 919, Zele
  - Boehringer Ingelheim Investigational Site 920, Zichem
  - Boehringer Ingelheim Investigational Site 921, Zichem
  - Boehringer Ingelheim Investigational Site 922, Zillebeke
  - Boehringer Ingelheim Investigational Site 923, Zonhoven
  - Boehringer Ingelheim Investigational Site 924, Zonnebeke
  - Boehringer Ingelheim Investigational Site 925, Zottegem
  - Boehringer Ingelheim Investigational Site 926, Zottegem
  - Boehringer Ingelheim Investigational Site 927, Zottegem
  - Boehringer Ingelheim Investigational Site 928, Zottegem
  - Boehringer Ingelheim Investigational Site 929, Zottegem
  - Boehringer Ingelheim Investigational Site 930, Zottegem
  - Boehringer Ingelheim Investigational Site 931, Zoutleeuw
  - Boehringer Ingelheim Investigational Site 932, Zoutleeuw
  - Boehringer Ingelheim Investigational Site 933, Zoutleeuw
  - Boehringer Ingelheim Investigational Site 934, Zoutleeuw
  - Boehringer Ingelheim Investigational Site 935, Zulte
  - Boehringer Ingelheim Investigational Site 936, Zwijnaarde

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 163 patients without information on albuminuria at baseline were enrolled to the study in addition. However, for these patients information on study completion is not available.
Period: Overall Study
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan
Started | 2027 (Baseline Population) | 684 (Baseline Population)
Completed | 1284 | 457
Not Completed | 743 | 227
Not completed — no respect of the 12 weeks period | 657 | 227
Not completed — Lost to Follow-up | 86 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for patients with available information on albuminuria at baseline. Respective data were not collected for patients without information on albuminuria at baseline.
Groups:
- Patients Without Albuminuria Treated With Telmisartan; Patients With Albuminuria Treated With Telmisartan: baseline population
- Total: Total of all reporting groups
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan | Total
Number analyzed (Participants) | 2027 | 684 | 2711
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11.7) | 65.9 (11.9) | 63.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 966 | 329 | 1295
  Male | 1061 | 355 | 1416

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Controlled Blood Pressure
Description: Systolic blood pressure (SBP) < 140 mmHg and diastolic blood pressure (DBP) < 90 mmHg if the patient has:
  * no chronic renal insufficiency or macroalbuminuria-dipsticks negative,
  * albuminuria is < 300 mg/24h or < 200 mg albumin per gram of creatinine
  * no diabetes
  or SBP < 130 mmHg and DBP < 80 mmHg if the patient has:
  * chronic renal insufficiency or macroalbuminuria-dipsticks are positive, albuminuria ≥ 300 mg/24h or ≥ 200 mg albumin per gram of creatinine
  * diabetes (type 1 or 2)
Time Frame: approximately 12 weeks (10 to 14 weeks) after baseline
Population: 1741 patients had a visit 2 between 10 and 14 weeks after baseline (1284+457)
Measure: Number; unit: Percentage of patients
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan
Number analyzed (Participants) | 1281 | 457
Percentage of patients | 46.1 (1.39) | 24.1 (2)
Statistical Analysis 1: Comparison: Patients Without Albuminuria Treated With Telmisartan vs Patients With Albuminuria Treated With Telmisartan; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Mean Difference in Systolic Blood Pressure
Description: The fall in systolic blood pressure (SBP) after approximately 12 weeks of treatment including telmisartan defined as SBP (baseline) - SBP (12 weeks) expressed in mmHg
Time Frame: baseline and approximately 12 weeks
Population: 1741 patients had a visit 2 between 10 and 14 weeks after baseline (1284+457)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan
Number analyzed (Participants) | 1281 | 457
mmHg | 20.8 (13.3) | 20.5 (13.0)

3. Secondary Outcome: Mean Difference in Diastolic Blood Pressure
Description: The fall in diastolic blood pressure (DBP) after approximately 12 weeks of treatment including telmisartan defined as DBP (baseline) - DBP (12 weeks) expressed in mmHg
Time Frame: baseline and approximately 12 weeks
Population: 1741 patients had a visit 2 between 10 and 14 weeks after baseline (1284+457)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan
Number analyzed (Participants) | 1281 | 457
mmHg | 11.7 (9.22) | 12.5 (8.53)

4. Secondary Outcome: Percentage of Patients With a Decrease of Systolic Blood Pressure (SBP) ≥ 10 mmHg (Responders)
Description: The response in SBP after approximately 12 weeks of treatment including telmisartan defined as a fall in SBP (SBP (baseline) - SBP (12 weeks) ≥ 10 mmHg
Time Frame: approximately 12 weeks (10 to 14 weeks) after baseline
Population: 1741 patients had a visit 2 between 10 and 14 weeks after baseline (1284+457)
Measure: Number; unit: Percentage of patients
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan
Number analyzed (Participants) | 1281 | 457
Percentage of patients | 87.7 (0.92) | 88.6 (1.49)

5. Secondary Outcome: Percentage of Patients Presenting an Adverse Event (AE)
Description: Percentage of patients with any adverse events during the study period, related or not to investigational drug
Time Frame: baseline to the end of study period
Population: 1741 patients had a visit 2 between 10 and 14 weeks after baseline (1284+457)
Measure: Number; unit: percentage of patients
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan
Number analyzed (Participants) | 1284 | 457
percentage of patients | 0.7 | 0.44

6. Secondary Outcome: Percentage of Patients With Positive to Negative Shift in Albuminuria
Description: Percentage of patients shifting from with (positive) albuminuria at baseline to without (negative) albuminuria after approximately 12 weeks
Time Frame: Approximately 12 weeks (10 to 14 weeks) after baseline
Population: All patients with albuminuria at initial visit and for which information on albuminuria was known at visit 2, 12 weeks after the initial visit.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Patients With Albuminuria Treated With Telmisartan
Number analyzed (Participants) | 331
Percentage of patients | 53.8 [48.4 to 59.2]

ADVERSE EVENTS:
Time Frame: From signing of informed consent through the end of the study
Description: 2874 participants at risk= patients without major protocol violation
Groups:
- EG002: patients without baseline albuminuria data
Arm/Group | Patients Without Albuminuria Treated With Telmisartan | Patients With Albuminuria Treated With Telmisartan | EG002
Serious Adverse Events (participants affected / at risk) | 1/2027 | 1/684 | 0/163
Other Adverse Events (participants affected / at risk) | 0/2027 | 0/684 | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Without Albuminuria Treated With Telmisartan (N=2027) | Patients With Albuminuria Treated With Telmisartan (N=684) | EG002 (N=163)
Ovarian metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myocardial infarct (Cardiac disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Observational study of daily medical practice, a lot of patients did not return to their GP for the second visit during the time period of 10 to 14 weeks after the first visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.